CLINICAL TRIAL: NCT00676624
Title: Infectious Causes of Uveitis, With Special Focus on Infection With Leptospira
Brief Title: Infectious Causes of Uveitis
Status: Completed | Type: Observational
Sponsor: Statens Serum Institut (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Steen Villumsen, MD, PhD, Statens Serum Institut
Other Study IDs: H-B-2007-097
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Uveitis
Keywords: uveitis; vitrectomy; infection; severe
MeSH Terms: conditions — Uveitis; Infections; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Corpus vitreum (vitreus body) Aqua from the anterior champer Whole blood in dry container Whole blood in container containing EDTA Whole blood in QuantiFERON test KIT for tuberculosis Urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Uveitis: Patients suffering from uveitis, who have vitrectomy performed for diagnostic purpose
- Control group: Patients suffering from either "Epiretinal fibrosis" og "Macula hole" who have vitrectomy performed for curative reasons

SUMMARY:
Uveitis is an inflammatory disease of one or both eyes. Uveitis will in severe cases lead to permanent loss of vision/blindness on the affected eye. Uveitis can be caused by autoimmune disease, infections and rarely trauma, but 50 % of the cases remain of unknown origin. Intraocular infections are from previous studies, known to be responsible for approximately 40 % of the cases of severe forms of uveitis. Most infectious causes of uveitis have the potential to be treated with antibiotic.

Most infectious causes of uveitis are under normal condition only possible to detect by using very specific detection methods. Further more it is often necessary to study a sample from with-in the eye (vitrectomy to get a proper diagnosis. The knowledge about witch kind of infections that causes uveitis, are therefore limited to the kind of infections that are tested for.

Our hypothesis are that infections are a frequent cause of severe uveitis in Denmark, and that by using a broad diagnostic approach it is possible to identify new or less recognized infections agents that are associated with uveitis. By this study we want to describe the prevalence and distribution of infections among patients with severe uveitis. In this study are we only including patients with a severe form of uveitis from a referral-hospital setting, where vitrectomy is done for a diagnostic purpose.

The patients will undergo a standard diagnostic examination including the most common infectious causes of uveitis. Beside this we will look for a broad range of infection, which has previously been described in the litera-ture to cause uveitis, but are not normally tested for. Further more, we will use broad ranged molecular diagnostic methods to look for new previously unknown bacterial causes of uveitis. Such study has not previously been done previously in Denmark. As control group are included patients that undergo vitrectomy for due either one of the two diseases "epiretinal fibrosis or "macula hole". All patients and controls will be interview using a standardized questionnaire about risk factors for acquiring these infections.

DETAILED DESCRIPTION:
All patients included eye examination that includes split-lamp examination with semi-quantification evaluation of the inflammation, fundoscopy incl. picture, and angiography.

Hemoglobin (Hb), Erythrocyte-volume fraction (EVF), Middle cell volume (MCV), middelcell hemoglobin concentration (MCHC), Trombocyte

* Alanin-aminotransferase (ALAT), S-albumin, S-bilirubin (total), Protrombin complex, INR.
* Na, K, creatinin,
* CRP, Leukocyte and differential count
* ACE (Angiotensin Converting Enzyme)
* S-Ca2+

X-ray of thorax

The biopsies taken from the patient are in the routine program are patients tested for intraocular infections with Herpes Simplex Virus, Cytomegalovirus, Varicella Zoster virus, Epstein-Barr virus and toxoplasma with PCR and serology on serum. Test for others infections like Candida spp. and Toxocare are done if clini-cally indicated. Other test includes cytopathological test of the corpus vitreum for cancer cells and serological test for Syphilis.

Beside the above mentioned test will we in this study test for:

Infections with Leptospira, Bartonella, Brucella, Mycobacterium tuberculosis, Leptospira, Toxocare, Borrelia, HIV.

We will use unspecific molecular test for Bacteria under a special setup to avoid DNA contamination. Culture of Leptospira will be done on urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Glostrup Hospital refferal eye clinic with uveitis were vitrectomy will be performed for diagnostic reasons

Exclusion Criteria:

* patients where eye surgery has been performed on the affected eye, within 30 days before the current vitrectomy
* Patients with known lymphoma
* Patient with clinical suspicion of intra-ocular cancer disease
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient at a referal hospital eye clinic with uveitis were vitrectomy will be performed for diagnostic reasons
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Prevalence and distribution of intraocular infections in the study group | September 2010

SECONDARY OUTCOMES:
The value of non-specific molecular diagnostic methods for detection of bacteria in the study group | September 2010

CONTACTS AND LOCATIONS:
Overall Officials: Steen Villumsen, MD PhD stud, Principal Investigator — Statens Serum Institut; Morten la Cour, MD DMSc, Study Chair — Glostrup University Hospital, Copenhagen; Karen A Krogfelt, Prof. PhD, Study Chair — Statens Serum Institut; Helle J Fuchs, MD, Study Chair — Glostrup University Hospital, Copenhagen; Jan U Prause, MD Prof DMSC, Study Chair — University of Copenhagen; Henrik V Nielsen, PhD, Study Chair — Statens Serum Institut; Lars P Nielsen, MD, Study Chair — Statens Serum Institut; Vibeke Thomsen, Cand Scient, Study Chair — Statens Serum Institut; Anne-Mette Lebech, MD, DMSc, Study Chair — Hvidovre University Hospital; Jorgen S Jensen, MD DMSc, Study Chair — Statens Serum Institut
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Denmark

REFERENCES:
- [Background] Bodaghi B, Cassoux N, Wechsler B, Hannouche D, Fardeau C, Papo T, Huong DL, Piette JC, LeHoang P. Chronic severe uveitis: etiology and visual outcome in 927 patients from a single center. Medicine (Baltimore). 2001 Jul;80(4):263-70. doi: 10.1097/00005792-200107000-00005. No abstract available. PMID 11470987